CLINICAL TRIAL: NCT06621212
Title: A Prospective, Multi-center, Phase 2 Study of Mitoxantrone Hydrochloride Liposome Injection Combined With Standard-dose Cytarabine and Venetoclax in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Mitoxantrone Hydrochloride Liposome, Standard-dose of Cytarabine and Venetoclax in the Treatment of R/R AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-AML-K16
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukaemia; Myeloid Malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAV regimen (Experimental): First induction: Mitoxantrone hydrochloride liposome injection, cytarabine combined with venetoclax.
  Second induction: Patients who achieved PR or MLFS after the first induction cycle will receive re-induction therapy with the same initial regimen.
  Consolidation: For patients with CR/CRi, allo-HSCT is recommended. For those currently ineligible for allo-HSCT, age- and fitness-adapted consolidation is advised. For intensive chemotherapy: Cytarabine (<60y: 2g/m² q12h d1-3; ≥60y: 1g/m² q12h d1-3) + Venetoclax 300mg d1-7, for 2-3 cycles. For non-intensive candidates, an appropriate regimen should be selected per investigator.
  Interventions: Drug: mitoxantrone hydrochloride liposome; Drug: Cytarabine; Drug: Venetoclax

INTERVENTIONS:
Drug: mitoxantrone hydrochloride liposome — Mitoxantrone hydrochloride liposome (30 mg/m^2) on day 1, every 4 weeks
Drug: Cytarabine — Cytarabine (100 mg/m^2 ) on day 1-7, every 4 weeks
Drug: Venetoclax — Venetoclax 100 mg on day 2，200 mg on day 3，400 mg on day 4-8, every 4 weeks

SUMMARY:
The purpose of this prospective, multi-center, single-arm, phase 2 study is to evaluate the efficacy and safety of a combination regimen of mitoxantrone hydrochloride liposome injection, standard-dose of cytarabine and venetoclax (MAV) in the treatment of relapsed or refractory (R/R) AML. The study plan to enroll 72 R/R AML patients who are expected to receive laboratory tests of bone marrow and blood specimens at regular times after MAV treatment.

DETAILED DESCRIPTION:
For patients with R/R AML, there is currently no established standard treatment. Previous research suggests that mitoxantrone could against venetoclax-resistant leukemia stem cells (LSCs) by modulating mitochondrial calcium levels. Based on the potentially synergistic killing effect of mitoxantrone and venetoclax, a phase 2 study is underway in R/R AML. Patients receive mitoxantrone hydrochloride liposome, moderate-dose of cytarabine (1.0 g/m^2, IV, q12h, d1, 3, 5) and venetoclax (MAV) when they were enrolled.

Here the investigator also conduct another phase 2 study of MAV regimen with standard-dose of cytarabine in relapsed or refractory (R/R) AML, aiming to evaluate the efficacy and safety of MAV regimen. All participants will receive MAV treatment including 30 mg/m^2 mitoxantrone hydrochloride liposome on day 1, 100 mg/m^2 cytarabine on days 1-7 and 400 mg venetoclax on days 2-8 with a dose escalation on days 2-4. Each cycle consists of 4 weeks. A maximum of 2 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
2. Age ≥18
3. Clinically diagnosed relapsed/refractory AML, excluding acute promyelocytic leukemia.

   1. Patients who failed after at least 1 courses of initial induction therapy.
   2. Bone marrow blasts≥5% after CR/CRi, or reappearance of blasts in the blood in at least 2 peripheral blood samples at least one week apart, or leukemia cell infiltration appeared in extramedullary.
   3. Conversion from MRD negativity to MRD positivity after CR/CRi.
4. Physical status score of Eastern Oncology Collaboration Group (ECOG) 0-2.
5. Life expectancy > 3 months.
6. AST/ALT≤2.5 ULN (for subjects with hepatic infiltration≤5 ULN); Total bilirubin≤1.5 ULN (for subjects with hepatic infiltration≤3 ULN); Serum creatinine≤1.5 ULN.

Exclusion Criteria:

1. Previous anti-tumor therapy meets one of the following criteria:

   1. Prior therapy with mitoxantrone or mitoxantrone liposome;
   2. Prior therapy with doxorubicin or anthracyclines, and the cumulative dose of doxorubicin > 360 mg/m^2 (1 mg doxorubicin was equivalent to 2 mg daunorubicin or 0.5 mg idarubicin);
   3. Have received other anti-tumor therapy (including chemotherapy, targeted therapy, hormone therapy, Chinese medicines with anti-tumor activity, except those that do not affect the efficacy of the study as determined by the investigator) or participated in other clinical trials and received clinical trial drugs within 4 weeks or 5 half-lives of the drug before the study;
2. Subjects who received strong or moderate CYP3A inducers/inhibitors or P-glycoprotein (P-gp) inhibitors within 7 days before starting study treatment;
3. Subjects who are unable to take oral medications or have malabsorption syndrome;
4. Cardiovascular diseases, including but not limited to:

   1. QTc interval >480 ms or long QTc syndrome in screening;
   2. Complete left bundle branch block, 2 or 3 grade atrioventricular block;
   3. Requiring treatment of serious and uncontrolled arrhythmia;
   4. New York Heart Association NYHA≥2;
   5. Cardiac ejection fraction (EF) was less than 50%;
   6. Myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other history of arrhythmia or clinically serious pericardial disease that requires treatment within the first 6 months of enrollment, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
5. Central nervous system leukemia;
6. Previous or current occurrence of other malignancies (in addition to non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years).
7. Subjects are suffering from any other uncontrollable disease (including but not limited to: uncontrolled diabetes and hypertension, and advanced infection);
8. HIV infection.
9. HBsAg or HBcAb positive, with HBV-DNA≥1x10^3 copies/mL; or HCV-RNA≥1x10^3 copies/mL;
10. A history of immediate or delayed allergy to similar drug and excipients of the investigate drug.
11. Pregnant, lactating female or subjects who refuse to use effective contraception during the study.
12. With a history of severe neurological or psychiatric illness.
13. Not suitable for this study as decided by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) rate | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Complete remission plus complete remission with incomplete hematologic recovery (CR+CRi). Response is assessed according to the the European LeukemiaNet (ELN) 2022 criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  CR+CRi+morphologic leukemia-free state+partial remission (CR+CRi+MLFS+PR). Response is assessed according to the the European LeukemiaNet (ELN) 2022 criteria.
Relapsed free survival (RFS) | up to 12 months
  Defined only for patients achieving CR or CRi. Measured from the date of achievement of remission until the date of hematologic relapse or death from any cause.
Event free survival (EFS) | up to 12 months
  Defined for all patients in the study. Measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first.
overall survival (OS) | up to 12 months
  Defined for all patients in the study. Measured from day 1 of treatment to the date of death from any cause.
Rate of CR/CRi without minimal residual disease | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Percentage of participants who achieve a CR MRD-/CRi MRD- as defined by investigators based on ELN 2022 criteria. MRD level is detected by flow cytometry and negtive MRD is defined as MRD value <0.1%.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From day 1 of treatment to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard which including hematologic and non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China